CLINICAL TRIAL: NCT00027001
Title: Qigong Therapy for Heart Device Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R21AT000291-01 (NIH)
Record Dates: First submitted 2001-11-15; First posted 2001-11-16 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-07

CONDITIONS: Depressive Disorder; Cardiac Diseases
Keywords: Qigong, exercise, circulatory assist devices
MeSH Terms: conditions — Depressive Disorder; Heart Diseases; Motor Activity | interventions — Qigong

INTERVENTIONS:
Behavioral: Aerobic and Resistance Exercises
Behavioral: Qigong

SUMMARY:
The goal of this study is to improve the overall physical health and quality of life of patients attached to mechanical heart devices while awaiting heart transplantation. Qigong, an ancient Chinese exercise that involves active participation of the individual in the form of meditation, breathing exercises and simple physical movements, is used in combination with a structured exercise program. We are testing the hypotheses that Qigong, in combination with a structured exercise program that combines aerobic and resistance training will improve the cardiovascular health and improve the quality of life of patients on mechanical heart devices. To test these hypotheses, we are measuring cardiovascular function and quality of life parameters in patients attached to mechanical heart devices who have participated in the exercise program and have practiced Qigong, and comparing these measures to patients who participated in the exercise program, but did not practice Qigong. Information gained from this research will serve as a basis from which the application of exercise training and Qigong can be applied to the treatment of other chronic diseases in which the physical conditioning and/or quality of life of individuals is compromised.

DETAILED DESCRIPTION:
The goal of this study is to improve the overall physical health and quality of life of patients attached to mechanical hearts or assist devices while awaiting heart transplantation. Qigong, an ancient Chinese exercise that involves active participation of the individual in the form of meditation, breathing exercises and simple physical movements, will be used as an adjunct to the therapies, including a structured exercise program, currently provided to these patients at the University of Arizona Health Sciences Center. Based on the results of studies that have demonstrated physiological and psychosocial benefits of structured exercise programs and the practice of qigong, the following hypotheses are proposed: 1) a structured exercise program that combines aerobic and resistance training will improve the cardiovascular health of patients on mechanical hearts and assist devices; these conditioning effects will be amplified by the practice of Qigong; 2) a structured exercise program that combines aerobic and resistance training will improve the quality of life of patients on mechanical hearts and assist devices; these conditioning effects will be amplified by the practice of Qigong; 3) improved quality of life and physical conditioning effected by the structured exercise program and Qigong will enhance quality of life and physical conditioning after cardiac transplantation. To test these hypotheses, the following specific aims will be accomplished: 1) obtain pilot data to evaluate alterations in specific measures of cardiovascular function and health in patients attached to mechanical heart or assist devices who have participated in a structured aerobic/resistance exercise program, with and without Qigong; 2) obtain pilot data to evaluate alterations in specific quality of life measures in patients attached to mechanical heart or assist devices who have participated in a structured aerobic/resistance exercise program, with and without Qigong; 3) as part of the clinical follow-up of these patients following heart transplantation, obtain pilot data to evaluate specific parameters of cardiovascular health and quality of life of individuals who were attached to mechanical heart or assist devices prior to receiving the transplant. Information gained from this research will serve as a basis from which the application of exercise training and Qigong can be applied to the treatment of other chronic disease states in which the physical conditioning and/or quality of life of individuals is compromised.

ELIGIBILITY:
The subjects of this study are patients who have been implanted with either a total artificial heart or ventricular assist device.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2000-09; Study Completion 2003-06

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arizona Health Sciences Center, Tucson, Arizona, United States